CLINICAL TRIAL: NCT04672343
Title: IPrognostic Impact of the Nutritional Status of Individuals Aged 70 Years and Older With SARS-CoV-2
Brief Title: Prognostic Impact of the Nutritional Status of Individuals Aged 70 Years and Older With SARS-CoV-2
Acronym: CodePRONUT
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: PUTOT AOIc 2020
Record Dates: First submitted 2020-12-16; First posted 2020-12-17 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: SARS-CoV-2
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — from D0 to hospital discharge
Other: Querying the INSEE database — Vital status at 3 months and 12 months

SUMMARY:
Mortality due to Covid-19 is much higher in the elderly. There are several reasons for the vulnerability of the elderly to the coronavirus: a less efficient immune system, underlying chronic conditions, less protected living conditions. They may also present a poor nutritional state and/or degraded metabolic reserves aggravating an underlying state of frailty. The prevalence of the risk of undernutrition in elderly patients with COVID-19 is high. The evolution of the nutritional status of people aged 70 years or older infected with SARS-Cov-2 is not yet well known. The prognosis of these patients could depend on their nutritional status at the time of the disease. In view of the lack of data, it would be interesting to compare the risk of mortality based on nutritional status in individuals with vs. those without COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 test positive (positive PCR test or evocative CT scan) or negative (with clinical suspicion of COVID, negative PCR test and non-evocative CT scan)
* Age ≥ 70 years old
* Hospitalization at Dijon University Hospital
* Person or legal representative has not stated their opposition to inclusion in the study after being informed

Exclusion Criteria:

* Person subject to a measure of judicial safeguard
* Non-affiliated or non-beneficiary of national health insurance

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Seniors with CoV-2-RASS
Sampling Method: Non-Probability Sample
Enrollment: 426 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
Death | to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France

REFERENCES:
- [Result] Putot A, Guyot C, Manckoundia P, Van Wymelbeke-Delannoy V. Association of body mass index with long-term outcomes in older adults hospitalized for COVID-19: an observational study. Sci Rep. 2024 Mar 29;14(1):7512. doi: 10.1038/s41598-024-58388-x. PMID 38553629